CLINICAL TRIAL: NCT02820714
Title: A Pilot Study of BLI801 Laxative in Adults Experiencing Non-Idiopathic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLI801-204
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BLI801 Laxative (Experimental): BLI801 oral laxative
  Interventions: Drug: BLI801 Laxative

INTERVENTIONS:
Drug: BLI801 Laxative — BLI801 Laxative

SUMMARY:
The objective of this study is to evaluate BLI801 laxative in adults experiencing non-idiopathic constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age
2. Taking medication known to cause constipation. This medication should remain stable throughout the study.
3. Constipated, defined by the following criteria: Fewer than 3 spontaneous defecations per week and at least one of the following symptoms for the previous 4 weeks:

   * Straining during > 25% of defecations
   * Lumpy or hard stools in > 25% of defecations
   * Sensation of incomplete evacuation for > 25% of defecations

   Onset of constipation must coincide with the instruction of treatment with a constipating medication
4. Otherwise in good health, as determined by physical exam and medical history
5. If female, and of child-bearing potential, is using an acceptable form of birth control
6. Negative urine pregnancy test at screening (visit 1), if applicable
7. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

1. Subjects whose constipation diagnosis and symptoms predate the initiation of treatment with the constipating medication.
2. Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
3. Subjects who have had major surgery 30 days before Visit 1; appendectomy or cholecystectomy 60 days before Visit 1; abdominal, pelvic, or retroperitoneal surgery 6 months before Visit 1; bariatric surgery or surgery to remove a segment of the GI tract at any time before Visit 1
4. Medical conditions associated with diarrhea, intermittent loose stools, or constipation, which could confound the interpretation of the results, eg, fecal incontinence or irritable bowel syndrome. Subjects with irritable bowel syndrome (IBS) that has been previously diagnosed by a physician prior to initiation of the constipating therapy and that meets the following criteria, are excluded:

   1. Absence of a structural or biochemical explanation for the abdominal pain symptom
   2. At least 12 weeks during a period of 12 months, of abdominal discomfort or pain with at least 2 of the following 3 features:

      * Relieved with defecation, and/or
      * Onset associated with a change in frequency of stool, and/or
      * Onset associated with a change in form of stool.
5. Subjects taking other prohibited concomitant medications.
6. Subjects who are pregnant or nursing, or intend to become pregnant during the study
7. Subjects of childbearing potential who refuse a pregnancy test
8. Subjects who are allergic to any BLI801 component
9. Active substance or alcohol use that, in the opinion of the investigator, could compromise patient's ability to comply with the study instructions.
10. Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
11. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
12. Subjects who withdraw consent at any time prior to completion of Visit 1 procedures
13. Subjects who have had a colonoscopy within 2 weeks of Visit 1 or are scheduled to have a colonoscopy during their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
% of subjects with treatment response | 4 weeks
  Greater than or equal to 3 spontaneous bowel movements per week for 2 out of 4 weeks

SECONDARY OUTCOMES:
% of subjects with treatment emergent adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (3):
- United States (3):
  - Braintree Research Site 1, Mobile, Alabama
  - Braintree Research Site 3, Bastrop, Louisiana
  - Braintree Research Site 2, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No